CLINICAL TRIAL: NCT03153800
Title: Autologous Bronchial Basal Cells Transplantation for Treatment of Chronic Respiratory Disease (CRD) Including Chronic Obstructive Pulmonary Disease (COPD), Bronchiectasis (BE) and Pulmonary Fibrosis (PF)
Brief Title: Autologous Bronchial Basal Cells Transplantation for Treatment of CRD Including COPD, BE and PF
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Regend Therapeutics (Industry)
Collaborators: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017042
Record Dates: First submitted 2017-05-10; First posted 2017-05-15 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Chronic Respiratory Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bronchial basal cells (Experimental)
  Interventions: Biological: bronchial basal cells

INTERVENTIONS:
Biological: bronchial basal cells — Transplantation of autologous bronchial basal cells by fiberoptic bronchoscopy.

SUMMARY:
Chronic respiratory diseases including chronic obstructive pulmonary disease (COPD), bronchiectasis (BE) or pulmonary fibrosis (PF) are usually not curable with damaged pulmonary structure and function. Bronchial basal cells are proved to regenerate bronchus and alveoli to repair the pulmonary injuries. In this study, we intend to perform an open, single-armed phase I clinical trial by transplantation of autologous bronchial basal cells on patients suffered from COPD, BE or PF. During the treatment, autologous bronchial basal cells, which were isolated from fiberoptic bronchoscopy and expanded in vitro, will be injected directly into lesions by fiberoptic bronchoscopy after careful characterization. In the following 6 months, the safety and efficacy of the treatment will be monitored by measuring the key clinical indicators.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with COPD, BE or PF according to the guideline;
* Clinically stable for more than 4 weeks;
* Tolerant to fiberoptic bronchoscopy test;
* Written informed consent signed.

Exclusion Criteria:

* Pregnant or lactating women;
* Patients positive for syphilis, HIV;
* Patients with malignant tumor;
* Patients with serious significant pulmonary infection and need anti-infection treatment;
* Patients with serious heart disease(NYHA class Ⅲ-Ⅳ);
* Patients with a history of abusing alcohol and illicit drug;
* Patients participated in other clinical trials in the past 3 months;
* Patients assessed as inappropriate to participate in this clinical trial by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-04-05 (Actual); Primary Completion 2021-04-04 (Estimated); Study Completion 2021-10-04 (Estimated)

PRIMARY OUTCOMES:
Forced expiratory volume in one second (FEV1) | 1-6 months
  One of the indicators in pulmonary function test, a marker to assess airway obstruction
Diffusion capacity of CO (DLCO) | 1-6 months
  One of the indicators in pulmonary function test, the extent to which oxygen passes from the air sacs of the lungs into the blood

SECONDARY OUTCOMES:
The ratio of forced expiratory volume in the first one second to the forced vital capacity (FEV1/FVC) | 1-6 months
  One of the indicators in pulmonary function test, representing the proportion of a person's vital capacity that they are able to expire in the first second of forced expiration to the full vital capacity
Maximum mid-expiratory flow (MMF) | 1-6 months
  One of the indicators in pulmonary function test, standing for maximal (mid-)expiratory flow and is the peak of expiratory flow as taken from the flow-volume curve and measured in liters per second
Maximum voluntary ventilation (MVV) | 1-6 months
  One of the indicators in pulmonary function test, measuring the maximum amount of air that can be inhaled and exhaled within one minute
Forced vital capacity (FVC) | 1-6 months
  One of the indicators in pulmonary function test, indicating the maximum amount of air a person can expel from the lungs after a maximum inhalation
6-minute-walk test (6MWT) | 1-6 months
  An indicator to evaluate the exercise function of patients with moderate or severe pulmonary heart diseases
Modified medical research council (MMRC) chronic dyspnea scale | 1-6 months
  An indicator to evaluate the level of dyspnea
St. George's respiratory questionnaire (SGRQ) scale | 1-6 months
  A questionnaire to assess life quality affected by the respiratory problems
Imaging of lung by high resolution computed tomography (HR-CT) | 1-6 months
  HR-CT images of lung will be analyzed to indicate the pulmonary structure.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hopsital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/25383540